CLINICAL TRIAL: NCT05003024
Title: Comparison of Train of Four, Tetanus 50 Hz and Tetanus 100 Hz Recovery Following Rocuronium Induced Neuromuscular Block Reversed by Sugamamdex
Brief Title: Comparison of Train of Four, Tetanus 50 and 100 Hz Recovery After Rocuronium Block Reversed by Sugammadex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DECURATOF
Record Dates: First submitted 2021-07-22; First posted 2021-08-12 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Residual Curarization
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOF scan train of four ratio monitoring (Active Comparator): Recovery of train of four ratio after sugammadex administration
  Interventions: Device: TOF SCAN
- ITF device tetanus stimulation monitoring (Experimental): Recovery of tetanus 100 Hz ratio after sugamamdex administration
  Interventions: Device: ITF

INTERVENTIONS:
Device: TOF SCAN — For each included patient, 2 monitorings (TOF Scan and ITF device) will be placed, one on each hand.
  Once 2 contractions of the adductor pollicis muscle will be observed on the TOF Scan side following train of four stimulation, 2 mg/kg sugammadex will be injected. Train of four ratio (delivered every minute) will be recorded.
  This sequence (tetanus 100 Hz followed by tetanus 50 Hz) will be repeated 5 times For each tetanus stimulation, the ratio between the residual force and the maximum force generated by the adductor pollicis muscle will be recorded (this ratio illustrates the fade phenomenon). At the end of this period lasting 23 minutes after sugammadex administration, anesthetic drug delivery will be stopped and the patient wil be allowed to recover.
  Arms: TOF scan train of four ratio monitoring
Device: ITF — For each included patient, 2 monitorings (TOF Scan and ITF device) will be placed, one on each hand.
  On the ITF device side, 3 minutes after sugammadex administration, a tetanus 100 Hz stimulation will be done followed 2 minutes later by a tetanus 50 Hz stimulation.
  This sequence (tetanus 100 Hz followed by tetanus 50 Hz) will be repeated 5 times For each tetanus stimulation, the ratio between the residual force and the maximum force generated by the adductor pollicis muscle will be recorded (this ratio illustrates the fade phenomenon). At the end of this period lasting 23 minutes after sugammadex administration, anesthetic drug delivery will be stopped and the patient wil be allowed to recover.
  Arms: ITF device tetanus stimulation monitoring

SUMMARY:
Despite neuromuscular transmission monitoring and pharmacological reversal allowing a train of four ratio recovery higher than 0.9, patients receiving neuromuscular blocking agent during general anesthesia have a high risk of postoperative pulmonary complications. While this train of four ratio thershold is considered as the gold standard to confirm the lack of residual paralysis, tetanus 100 Hz stimulation showed a marked fade. This result has been observed in absence of reversal agent administration.

Therefore, the present study has been designed to compare the recovery of train of four stimulation, tetanus 50 Hz and tetanus 100 Hz stimulation in patient receiving rocuronium during general anesthesia and reversed by a specific reversal agent (sugammadex). The sugammedex will be injected once two muscular contractions of the adductor pollicis muscle will be observed after a train of four stimulation, at a dose (2mg/kg) in accordance with the clinical practice worldwide admitted.

Two questions have to be investigated. First, is this dose of sugammadex sufficient to allow a complete recovery of tetanus stimulations? Second, due to the pharmacological properties of sugammadex, does a recurarisation phenomenon occur following repeated tetanus stimulations? The attented results of this study will be to propose a new thinking on what we really need to make relevant progress in the safety aspects of residual paralysis outcome.

ELIGIBILITY:
Inclusion Criteria:

* ASA clinical status 1 to 3
* Informed consent obtained before anesthesia induction

Exclusion Criteria:

* ASA clinical status 4
* Emergency surgery; scheduled surgery in prone position,
* Hepatic or renal disease,
* BMI higher than 35,
* Allergy to rocuronium or sugammadex

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
To compare the recovery of train of four ratio with the tetanus 100 Hz ratio following sugammadex administration to reverse the rocuronium induced neuromuscular bock at the end of the surgical procedure | 23 minutes after sugammadex administration
  delay following sugammadex administration to obtain a train of four ratio higher than 0.9 and a tetanus 100 Hz ratio higher than 0.9

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No